CLINICAL TRIAL: NCT05349344
Title: Effect of Aerobic Exercise Training on Premenstrual Syndrome Symptoms and Health Related Quality of Life Among Working Women
Brief Title: Effect of Aerobic Exercise on Premenstrual Syndrome Symptoms (PMS).
Acronym: PMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/00841 Hareem Javed
Record Dates: First submitted 2021-08-11; First posted 2022-04-27 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Premenstrual Syndrome; Quality of Life
Keywords: Aerobic Training
MeSH Terms: conditions — Premenstrual Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aerobic Circuit Training (Experimental): Each session consists of 5 minutes of warming up,20 minutes of aerobic exercises with brief resting periods, followed by 5 minutes to cool down.
  Interventions: Other: Aerobic circuit training
- outdoor walk (Active Comparator): 30minutes Walking outside below 40% of HR max for 2 months.(3 times per week for 8 weeks).
  Interventions: Other: Outdoor walk

INTERVENTIONS:
Other: Aerobic circuit training — Aerobic Exercise Training, 3 times a week for 8 weeks, (Tuesday, Thursday & Saturday, 24 sessions Total) 30 min each time, at 60-80 % of HR max (moderate intensity).
  Arms: Aerobic Circuit Training
Other: Outdoor walk — 30minutes Walking outside below 40% of HR max for 2 months.(3 times per week for 8 weeks).
  Arms: outdoor walk

SUMMARY:
To Determine the Effect of Regular Aerobic Exercise Training on Severity of Premenstrual Syndrome Symptoms and Health-Related Quality of life on working women.Exercise can be used as an alternative therapy in reducing premenstrual symptoms.But still there is lack of Literature on PMS in work Place and effect of Treatments to improve overall Quality of life in working women.And this study aims to fill the gap by assessing the impact that Premenstrual Syndrome can have on working women's Quality of life and can be used to establish a model of regular exercise program with the potential to decrease premenstrual symptoms and improve quality of life for a menstrual health-friendly workplace environment for Female Employees.

DETAILED DESCRIPTION:
A review conducted to assess the effect of 8 weeks of aerobic exercise on the non-athletic females facing premenstrual syndrome symptoms. The results displayed positive effects of 8 weeks of exercise on symptoms of PMS. The aerobic exercise helped to reduce both psychological and physical symptoms.

Regular swimming for 8 weeks also decreased the severity of PMS symptoms in females. Results deduced that the exercise improved the vascular activity of the heart, and reduced stress and anxiety. Moreover, it also enhanced bone density.

In one of RCT the effect of 3 months of exercise through treadmill on PMS and hormones was also evaluated. It was assumed that many symptoms of PMS were reduced including the carbohydrate cravings, stress, and depression. The electrolyte change was also reduced. Exercise also reduced the proportion of backache and menstrual cramps in females.

Another review on a balanced diet and regular exercise demonstrated that the diet rich in the essential nutrients and regular exercise improved the health of the females. The symptoms of PMS were also reduced in these females along with the intensity of dysmenorrhea.

ELIGIBILITY:
Inclusion Criteria:

* Regular menstrual cycles (cycles of 21-35days with a bleeding time of 3-10days).
* PMS (as per screening questionnaire PSST Criteria).
* No history of psychiatric disorder (Score below 40 from Beck Depression questionnaire).
* Women working in hospital settings (health care Professionals).

Exclusion Criteria:

* No history of co-existing Medical illness including DM, Thyroid dysfunction, Hypoglycemia, Cardiac Pathologies.
* Women undergone Hysterectomy or other Gynecological procedure.
* Women on medications i.e. Contraceptive pills and HRT.
* Pregnant women.
* History of drug abuse or Alcohol intake.
* Participation in another sports program

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Reproductive aged working women.
Enrollment: 50 (Actual)
Dates: Start 2020-09-20 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
Severity of Premenstrual Syndrome Symptoms. Premenstrual Syndrome Scale (PMSS) | 8 weeks
  Use to Assess severity of Premenstrual Syndrome Symptoms. This Instrument has 40 questions with three sub-scales(Physiological,Psychological and Behavioral symptoms).
  It has 5-point Likert-style scale.

SECONDARY OUTCOMES:
Effect on Health- Related Quality of Life. | 8 weeks
  Use to Assess Health-Related Quality of Life. It consists of five questions,and Likert -type, Measurements of scale are set according to as a range from one (none of the time) to five (all of the time).

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Ehsan, PP-DPT, Principal Investigator — Riphah International University
Locations (1):
- Fauji Foundation hospital, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Maged AM, Abbassy AH, Sakr HRS, Elsawah H, Wagih H, Ogila AI, Kotb A. Effect of swimming exercise on premenstrual syndrome. Arch Gynecol Obstet. 2018 Apr;297(4):951-959. doi: 10.1007/s00404-018-4664-1. Epub 2018 Jan 19. PMID 29350276
- [Background] El-Lithy A, El-Mazny A, Sabbour A, El-Deeb A. Effect of aerobic exercise on premenstrual symptoms, haematological and hormonal parameters in young women. J Obstet Gynaecol. 2015 May;35(4):389-92. doi: 10.3109/01443615.2014.960823. Epub 2014 Oct 3. PMID 25279689
- [Background] Yilmaz-Akyuz E, Aydin-Kartal Y. The effect of diet and aerobic exercise on PremenstrualSyndrome: Randomized controlled trial. Revista de Nutrição. 2019;32